CLINICAL TRIAL: NCT01155492
Title: Increased Gut Permeability to Lipopolysaccharides (LPS) in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Kathleen M. Shannon, Professor, Neurological Sciences, Rush University Medical Center
Other Study IDs: 07100403
Record Dates: First submitted 2010-06-15; First posted 2010-07-01 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Parkinson's Disease; Multiple System Atrophy
Keywords: lipopolysaccharides; etiology; inflammation; colonic bacteria; intestinal permeability
MeSH Terms: conditions — Parkinson Disease; Multiple System Atrophy; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Colonic mucosa biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Subjects with Parkinson's disease: Male and female subjects with clinically diagnosed Parkinson's disease, Stage I-IV.
- Control subjects: Age- and gender-matched subjects who do not have Parkinson's disease
- Multiple system atrophy.: Men and women with clinically diagnosed multiple system atrophy.

SUMMARY:
The gut may be a portal of entry for agents that cause or contribute to the causes of Parkinson's disease (PD). The investigators are studying changes in the normal population of gut flora and in intestinal permeability and their associations with early PD.

DETAILED DESCRIPTION:
Clinical and pathological data suggest Parkinson's disease (PD) may result from an inflammatory process beginning in the intestinal wall that initiates alpha-synuclein aggregation, which then spreads from neuron to neuron, reaching the central nervous system. Bacteria living within the intestinal tract produce lipopolysaccharide endotoxin, a toxin known to induce parkinsonism in animal models. We hypothesize that exposure to LPS, either from excessive production or excessive absorption may be the cause of this inflammation. This study aims to: (1) describe differences in the population of gut bacteria in PD compared to control subjects; (2) assess leakiness of the gut wall by differential absorption of non-absorbable sugars; (3) measure plasma levels of endotoxin and inflammation; and (4) study characteristic PD pathology and evidence of inflammation in biopsy samples of the colon obtained by sigmoidoscopy.

ELIGIBILITY:
Inclusion Criteria--Parkinson's disease:

* Clinically diagnosed Parkinson's disease
* Hoehn & Yahr stage 1-2.5
* No symptomatic treatment of Parkinson's disease symptoms

Inclusion Criteria--Multiple System Atrophy

* Clinically diagnosed Multiple System Atrophy.

Inclusion Criteria--Control subjects:

* No diagnosis of Parkinson's disease and no signs of Parkinson's disease on screening neurological examination

Exclusion Criteria:

* Secondary or atypical parkinsonism other than Multiple System Atrophy
* Occupation or medical treatment known to influence intestinal flora
* Organic gastrointestinal disease other than hiatal hernia or hemorrhoids; history of gastrointestinal surgery other than remote appendectomy or cholecystectomy.
* Acute or chronic medical illness that would confound study results.
* Coagulopathy or use of anticoagulant medications (including aspirin).
* Chronic use of diuretics

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with Parkinson's disease Age- and gender-matched controls
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2007-09; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Total urine sugar per 24 hours | 24 hours
  Subjects consume a mixture of sugars (lactulose, sucrose), then collect urine for 24 hours. Sugar concentrations in the urine are assayed by gas chromatography.
LH-PCR fingerprint analysis | 24 hours
  Total genomic DNA will be extracted from colonic mucosa biopsy specimens and lumenal samples, and will be amplified by PCR using bacterial primers. PCR products will be separated and analyzed for amplicon length heterogeneity.
Blood endotoxin and cytokine levels | 24 hours
  Blood endotoxin and cytokine levels
Histopathology and immunohistochemistry of colonic mucosa | 24 hours
  A portion of the colonic tissue will be studied with histopathology and immunohistochemistry techniques for alpha-synuclein pathology, cytokines and inflammatory markers.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Shannon, M.D., Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Forsyth CB, Shannon KM, Kordower JH, Voigt RM, Shaikh M, Jaglin JA, Estes JD, Dodiya HB, Keshavarzian A. Increased intestinal permeability correlates with sigmoid mucosa alpha-synuclein staining and endotoxin exposure markers in early Parkinson's disease. PLoS One. 2011;6(12):e28032. doi: 10.1371/journal.pone.0028032. Epub 2011 Dec 1. PMID 22145021